CLINICAL TRIAL: NCT00949741
Title: Observational Retrospective Multicenter Study for the Citofluorimetric Analysis of Cerebrospinal Fluid Vs Conventional Method in Patients With Aggressive Non-Hodgkin's Lymphoma Without Leptomeningeal Disease
Brief Title: Observational Study for the Cytofluorimetric Analysis of Cerebrospinal Fluid in Non-Hodgkin's Lymphoma Patients
Acronym: CFM
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Multiregionale per lo studio dei Linfomi e delle Leucemie (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Other Study IDs: CFM
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2009-07

CONDITIONS: Diffuse Large Cell Lymphoma; Lymphoblastic Lymphoma; Burkitt's Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to define if flow cytometry has more sensitivity for detecting neoplastic cells in cerebrospinal fluid versus conventional cytology.

DETAILED DESCRIPTION:
Aggressive B-cell non-Hodgkin's lymphoma (B-NHL), Lymphoblastic Lymphoma and Burkitt's Lymphoma are at high risk of CNS relapse. For this reason is recommended a prophylaxis therapy. This suggests that negative leptomeningeal localization patients at diagnosis are really positive and that would be a very high risk of CNS relapse subtype patients. It's very important detecting neoplastic cells in cerebrospinal fluid as soon as possible. This study will evaluate only patients that have been flow cytometry and cytology at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of

   * Diffuse large cell lymphoma HIV positive,
   * Lymphoblastic lymphoma,
   * Burkitt's lymphoma,
   * Mantle cell lymphoma blastoid type.
2. DLCL patients who presented one risk factor for leptomeningeal involvement as:

   * testis, bone marrow, orbit, palate, paranasal cavity or peridural disease localization,
   * 2-3 age-adjusted IPI score with more than 1 extranodal site and LDH > normal.
3. Patients with cytologic and flow cytometry on cerebrospinal fluid at diagnosis.

Exclusion Criteria:

1. Patients with clinical or strumental evidence of meningeal localization disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by aggressive non-Hodgkin's lymphoma at diagnosis
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of diagnostic agreement of citofluorimentria flow in the research of lymphoma cells in the cerebrospinal fluid vs cell morphology. | Evaluation at diagnosis
  Evaluation of diagnostic agreement of citofluorimentria flow in the research of lymphoma cells in the cerebrospinal fluid vs cell morphology. The second test will be performed independently and without the cytologist is aware of the outcome of the analysis by flow cytometry.

SECONDARY OUTCOMES:
Collection of all paper forms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Principal Investigator — SCDO Ematologia AOU San Giovanni Battista Torino Italy
Locations (12):
- Italy (12):
  - ASO SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - PO Centro Binaghi Divisione di Ematologia CTMO, Cagliari, CA
  - Az. Ospedaliero Universitaria Careggi, Florence, FI
  - Ospedale Vito Fazzi Divisione di Ematologia, Lecce, LE
  - Ospedale Cardinale Panico, Tricase, LE
  - IRCCS San Raffaele, Milan, MI
  - Ospedale San Gerardo, Monza, MI
  - Centro di riferimento Oncologico Divisione Oncologia A, Aviano, PN
  - AO Univ. Policlinico Tor Vergata Divisione di Ematologia, Roma, RM
  - Università La Sapienza Policlinico Umberto I, Roma, RM
  - Ematologia Università del Piemonte Orientalr, Novara
  - SCDO Ematologia 2 AOU San Giovanni Battista, Torino